CLINICAL TRIAL: NCT02990299
Title: mHealth for Diabetes Adherence Support
Acronym: mDAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Ben Gerber, Professor of Medicine, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2016-0380; 1R01DK108141 (NIH)
Record Dates: First submitted 2016-12-05; First posted 2016-12-13 (Estimated); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus, Type 2; Medication Adherence; Telemedicine; Community Health Workers; Pharmacists; Mobile Health
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Medication Adherence | interventions — Telemedicine

STUDY DESIGN:
Intervention Model Description: A 2-arm, parallel, randomized controlled trial. Patients are randomized 1:1 to (1) mHealth diabetes adherence support intervention for one year and monitored with usual care for the second year, or (2) wait-list usual care for one year, then intervention during the second year.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Participants will receive their usual care for the first year of their enrollment in the study. They will receive a referral to a diabetes educator and a clinical pharmacist, a one-page sheet of contact information for their healthcare providers, and paper-based, low-literacy diabetes information. After one year, they will change to the mDAS intervention arm for one year.
- mHealth for Diabetes Adherence Support (Experimental): Participants will receive in-person support from a health coach and a clinical pharmacist with whom they will meet with regularly via videoconference. After one year, participants who have completed the mDAS intervention will be monitored for an additional year with usual care to evaluate maintenance.
  Interventions: Behavioral: mHealth for Diabetes Adherence Support

INTERVENTIONS:
Behavioral: mHealth for Diabetes Adherence Support — Participants will be paired with a health coach who will provide ongoing support and resources in medication and lifestyle adherence and diabetes self-management. The health coach will perform regular home visits, telephone support and tailored text-messages based on the participant's preferences and needs. They will help assess barriers to adherence and use motivational interviewing to help patients set goals and create action plans. They will also facilitate videoconferences with an assigned clinical pharmacist who will provide consultation on medication use, reconciliation and adherence, identify therapeutic goals and formulate an approved plan of care.
  Other Names: mDAS
  Arms: mHealth for Diabetes Adherence Support

SUMMARY:
The purpose of this research study is to determine the benefit and cost of including health coaches, clinical pharmacists and mobile health (mHealth) tools such as text messaging and videoconferencing in diabetes management support services for African-Americans and Latinos with uncontrolled Type 2 Diabetes.

DETAILED DESCRIPTION:
Many African-Americans and Latinos with diabetes do not achieve recommended diabetes goals placing them at high risk for complications. Team-based models of care can help in reaching goals of therapy. Additionally, mobile health (mHealth) technologies can further improve outcomes among those more difficult to reach. This study will evaluate the impact of a team-based, mHealth intervention designed to improve medication adherence, healthy eating, and physical activity behaviors. The investigators will compare this mHealth approach with usual care.

Clinical pharmacists and health coaches (HC) will deliver our proposed team-based intervention. mHealth delivery includes mobile phone text messaging, secure videoconferencing, and HC home visits. Pharmacists will focus on medication reconciliation and adherence. Health coaches will help identify psychosocial and environmental challenges to adherence in a culturally-sensitive manner. Together, they can assist in goal-setting, problem-solving, negotiation of competing priorities, and provide social support leveraging mHealth technologies.

Preliminary data from previous research by the research team supports the role of health coaches partnering with clinic- based pharmacists in improving diabetes outcomes in minorities. In the proposed mHealth intervention, patient- pharmacist videoconferencing will eliminate the need for in-person visits with a pharmacist, which is impractical for many low-income patients. In addition, pilot work suggests that text messaging is a preferable means of communication and may facilitate more frequent contact with patients.

This is a randomized, controlled trial to evaluate the effectiveness of an mHealth diabetes adherence support intervention delivered by clinical pharmacists and health coaches. The research team will randomize 220 patients through UI Health to either: (1) mHealth diabetes adherence support through clinical pharmacists and health coaches; or (2) usual care. After one year, patients completing the mHealth intervention will be monitored for an additional year while the usual care group receives the mHealth approach. Outcomes include medication adherence, hemoglobin A1c, blood pressure, and LDL-cholesterol levels. The specific aims include: (1) evaluate the effectiveness of an mHealth diabetes adherence support intervention delivered by clinical pharmacists and health coaches to African-American and Latino adults with uncontrolled type 2 diabetes; (2) evaluate the maintenance of improved diabetes behaviors as well as clinical outcomes one year after completing the intervention; (3) evaluate the cost and cost-effectiveness of mHealth diabetes adherence support compared to usual care; and (4) evaluate the reach, adoption, and implementation of mHealth diabetes adherence support based on the RE-AIM framework.

ELIGIBILITY:
Inclusion Criteria:

* Self-identified as Latino/Hispanic or African-American
* Verbal fluency in English or Spanish
* Latest A1c ≥ 8.0% (within 3 mo)
* History of Type 2 Diabetes (> 1 year)
* Between the ages of 21 and 75 years
* Unlimited mobile phone/text messaging plan with ability to reply to text messages
* Home environment capable of video conferencing with wireless signal
* Receives primary care at UI Health clinical site for at least one year, with one visit during past year
* Able and willing to provide informed consent (agree to data collection requirements, accept randomization, agree to home visitation with HC and pharmacist involvement, and participate for two years)

Exclusion Criteria:

* Unable to verbalize comprehension of study or impaired decision making
* Family/household member already participating in same study
* Currently receiving regular pharmacist support through Medication Therapy Management or equivalent
* History of, or planned, gastric bypass or transplant surgery
* History of bipolar or psychotic disorder
* Other severe comorbidities that require complex, aggressive, or palliative treatment, e.g., stage 4 or greater renal disease, liver failure, cancer (other than nonmelanoma skin cancer), terminal illness
* Investigator discretion for safety concerns

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2017-03-24 (Actual); Primary Completion 2022-01-07 (Actual); Study Completion 2022-01-07 (Actual)

PRIMARY OUTCOMES:
Hemoglobin A1c | 24 months

SECONDARY OUTCOMES:
Self-reported medication adherence | 24 months
  A 3-item questionnaire will be administered to measure adherence to diabetes medications.
Blood Pressure | 24 months
LDL Cholesterol | 24 months
  LDL Cholesterol will be measured as part of a Full Lipid profile blood test.
Diabetes Self-Management | 24 months
  Self-management will be measured by the revised 11-item Summary of Diabetes Self Care Activities questionnaire.
Health related quality of life | 24 months
  General health-related quality of life will be measured by the EuroQOL 5D (EQ-5D).
Diabetes related quality of life | 24 months
  Diabetes-related quality of life will be measured by the Diabetes Distress Screening Instrument (DDS4).
Depression | 24 months
  Measured with the nine-item Patient Health Questionnaire (PHQ-9)
Alcohol Misuse | 24 months
  Measured using the 3-item AUDIT-C questionnaire
BMI | 24 months
  Height and weight will be taken at each time point to determine BMI
Social Support | 24 months
  4-item questionnaire measuring satisfaction with support from friends, family and health care team
Diabetes Self-efficacy | 24 months
  8 -item questionnaire measuring confidence in diabetes self-management skills

OTHER OUTCOMES:
Healthcare utilization | 24 months
  This will include costs associated with hospital admissions, emergency room and outpatient visits and prescription medications.
Program cost | 24 months
  This will include costs associated with the intervention including pharmacists and health coaches (training, salaries, implementation), educational materials, tablet computers and associated data service, text messaging and videoconferencing.
Health Coach Satisfaction | 1 year after health coach assignment
  A survey administered to the patient for feedback on their assigned health coach.

CONTACTS AND LOCATIONS:
Overall Officials: Ben S Gerber, MD, MPH, Principal Investigator — University of Illinois at Chicago; Lisa K Sharp, PhD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois Hospital and Health Sciences System, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sharp LK, Biggers A, Perez R, Henkins J, Tilton J, Gerber BS. A Pharmacist and Health Coach-Delivered Mobile Health Intervention for Type 2 Diabetes: Protocol for a Randomized Controlled Crossover Study. JMIR Res Protoc. 2021 Mar 10;10(3):e17170. doi: 10.2196/17170. PMID 33688847
- [Derived] Gerber BS, Biggers A, Tilton JJ, Smith Marsh DE, Lane R, Mihailescu D, Lee J, Sharp LK. Mobile Health Intervention in Patients With Type 2 Diabetes: A Randomized Clinical Trial. JAMA Netw Open. 2023 Sep 5;6(9):e2333629. doi: 10.1001/jamanetworkopen.2023.33629. PMID 37773498